CLINICAL TRIAL: NCT04974983
Title: Impact of Bevacizumab on Symptom Burden and Neurological Deficits in Patients With Recurrent GBM: A Retrospective Patient Chart Review
Brief Title: Impact of Bevacizumab on Symptom Burden and Neurological Deficits in Patients With Recurrent Glioblastoma
Status: Completed | Type: Observational
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Martin Proescholdt, Professor of Neurosurgery, University Hospital Regensburg
Other Study IDs: Z-2017-0901-5
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Glioblastoma; Angiogenesis
Keywords: Glioblastoma; Angiogenesis
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Treatment without bevacizumab
  Interventions: Other: Observation of neurological deficits
- B: Treatment with bevacizumab
  Interventions: Other: Observation of neurological deficits

INTERVENTIONS:
Other: Observation of neurological deficits — Observation of neurological deficits

SUMMARY:
This retrospective non - interventional patient chart review will be utilizing real world clinical data from patients treated for rGBM at the University Regensburg Medical center either with or without bevacizumab. Only patients will be analyzed who were potentially eligible for bevacizumab treatment. The study is designed to investigate the potential effects of bevacizumab treatment on the functional status, symptom burden, neurological deficits, time to tumor progression and overall survival between cohorts potentially eligible for bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of recurrent glioblastoma

Exclusion Criteria:

Severe neurocognitive deficits

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent glioblastoma either treated with or without bevacizumab
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Functional outcome | 15 months
  Neurological deficits impacting functional independency

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No